CLINICAL TRIAL: NCT06976931
Title: A Dose-escalation Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of YY2201 in Patients With Advanced Solid Tumors
Brief Title: Study on the Safe Dosage and Therapeutic Effect of the Drug YY2201 Tablets on Patients With Advanced Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jiangsu YaYao Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2504318-15
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study on the safe dosage and therapeutic effect of YY2201 tablets in patients with advanced cancer (Experimental)
  Interventions: Drug: YY2201

INTERVENTIONS:
Drug: YY2201 — This is a multicenter, open-label, dose-escalation phase I study. participants will receive one single target dose of YY2201 on Cycle 0 Day 1 (C0D1) to observe safety and collect PK blood samples up to 48 h post-dose. On the third day after the first dose (Cycle 1 Day 1, C1D1), subjects will start to receive multiple doses of YY2201 orally twice daily (approximately 12 h interval) for 3 days followed by 4 days off in a 21-days treatment cycle.

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of YY2201 in participants with advanced solid tumors. The main questions it aims to answer are:

What medical problems do participants have when taking drug YY2201? What is the maximum tolerated dose (MTD) in patients with advanced solid tumors? What is the anti-tumor efficacy of YY2201 in patients with advanced solid tumors This is a multicenter, open-label, dose-escalation phase I study.

Participants will:

Start to receive multiple doses of YY2201 orally twice daily (approximately 12 h interval) for 3 days followed by 4 days off in a 21-days treatment cycle Perform radiography tumor assessments at screening visit every 2 cycles. Keep a diary of their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntary to participate in the clinical study, sign a written ICF, and able to comply with clinical visits and study-related procedures.

  2.Male or female with age ≥18 when signing the ICF. 3.Has a histologically or cytologically confirmed advanced solid tumors who are refractory to or intolerant of available standard-of-care therapy or have no effective standard treatment available.

  4.ECOG performance score of 0 or1. 5.Expected survival of at least 3 months. 6.Adequate organ function (without any supportive treatment including blood components, growth factors, etc. within 7 days prior to the laboratory test): Bone marrow: neutrophil count (ANC) ≥ 1.5×109/L, platelet count (PLT) ≥ 90×109/L, and hemoglobin (HGB) > 9.0 g/dL.

Coagulation function: international normalized ratio (INR) and activated partial prothrombin time (APTT) prolonged to ≤1.5×ULN.

Liver function: total bilirubin (TBIL) ≤ 1.5×ULN or ≤ 3 × ULN in case of known Gilbert disease, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5×ULN, if there is liver metastasis, ALT or AST ≤ 5×ULN.

Renal function: creatinine clearance ≥ 60 mL/min (using Cockcroft-Gault formula).

Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%. 7.At least one measurable lesion according to the RECIST v1.1 criteria. 8.Eligible patients with fertility (male and female) must agree to use reliable contraceptive methods (hormonal or barrier method) with their partners during the trial period and at least 3 months after the last administration; female patients of childbearing age must have a negative serum pregnancy test within 7 days before the first dose of YY2201.

Exclusion Criteria:

* 1.Has received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immune checkpoint inhibitor therapy, other anti-tumor treatments, or other un-marketed investigational drugs within 4 weeks prior to first dose of YY2201 (or within 5 half-lives of treatment, whichever is shorter), except for the following items: Have used nitrosourea or Mitomycin C within 6 weeks prior to first dose of Y2201.

Have used oral fluorouracil and small molecule targeted drugs within 2 weeks or 5 half-lives of the drugs prior to first dose of YY2201 (whichever is longer).

Have used herbal therapy with anti-tumor indications are within 2 weeks prior to first dose of YY2201.

2.Has prior (within 2 years before screening) or concurrent other malignancy (except for cured basal cell carcinoma of the skin, carcinoma in situs of cervix, ductal carcinoma in-situ, and prostate cancer which not requiring treatment).

3.Has undergone major organ surgery (excluding biopsy) or have had significant trauma within 4 weeks prior to first dose of YY2201 or required elective surgery during the study period.

4.Is taking (or cannot be stopped at least 1 week prior to first dose of YY2201) any drug that is known to strongly or moderately inhibit or induce CYP2C8 and CYP3A4.

5.The adverse reactions of previous anti-tumor treatments have not yet recovered to grade ≤1 (except for toxicity judged by the investigator to have no safety risk, such as alopecia and fantigue).

6.Has spinal cord compression or brain metastases and requiring corticosteroid therapy at a dose of more than 10 mg prednisone or equivalent per day for at least 4 consecutive weeks prior to initiation of study treatment (unless asymptomatic, treated, and stable) or a history of leptomeningeal metastases.

7.Any gastrointestinal tract related conditions that may affect the drug absorption as judged by the investigator, such as nausea and vomiting that are difficult to control, intestinal obstruction, gastric outlet obstruction, unable to swallow preparations, previous major gastrointestinal resection and so on.

8.Has active infection 1 week before the first dose of YY2201 and currently need systemic anti-infection treatment.

9.HIV infection, or active HBV infection or active HCV infection, with the exception:

1. Patients with serologic evidence of chronic HBV infection and have HBV viral load below the limit of quantification with normal liver function.
2. Patients with serologic evidence of HCV infection and have negative hepatitis C virus RNA test results.

   10.History of serious cardiovascular and cerebrovascular diseases, including but not limited to: Severe cardiac rhythm or conduction abnormality, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrioventricular block, etc., PR interval > 250 ms; Thromboembolic events requiring therapeutic anticoagulation, or subjects with a venous filter; Patients with Class III~IV cardiac insufficiency according to the criteria of New York Heart Association (NYHA); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or higher cardiovascular and cerebrovascular events within 12 months prior to the first dose; QT interval corrected through Fridericia's formula (QTcF) prolongation (male > 450 ms, female > 470 ms); any factors that increase the risk of QTc prolongation and arrhythmia, such as heart failure, congenital long QT syndrome, family history of long QT syndrome, and QT interval prolongation caused by any concomitant drug.

   11.History of non-infectious pneumonitis (NIP)/pneumonitis requiring systemic steroids, or active NIP/ pneumonitis, or other severe lung disease.

   12.Substance use disorder that may interfere with the participant's involvement in the study or evaluation of the study result, as determined by the investigator.

   13.Patient with mental disorders, severe cognitive disorder, poor compliance, or is not suitable for participating in this clinical study determined by the Investigator.

   14.Women who are pregnant or breastfeeding. 15.Patient who cannot tolerate venous blood sampling. 16.Known allergy to YY2201 or any of its excipient. 17.History of other serious systemic diseases, or not suitable to participate in this study for other reasons as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2027-04-05 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) and Dose-limiting toxicity (DLT) events by the National Cancer Institute Common Terminology Criteria (CTCAE) version 5.0. | C0D1, C0D2, C1D1, C1D3, C1D8, C1D15, C1D17, C1D21, C2D1, C2D15, C3D1, C3D15, CnD1 (from C4), EOT+7 days and 28±7 days after the last dose of YY2201.（C=cycle,D=day,each cycle is 21 days）
  Electrocardiogram：12-lead ECG machine，heart rate(times/minute)； laboratory tests：blood cell analyzer(% of blood cells)，Chemistry Analyzer(Concentration of...)，Urine Analyzer(Rate of...),etc.